CLINICAL TRIAL: NCT03527706
Title: PREDICtors for Health Related Quality of Life After Elective Sigmoidectomy for DIVerticular Disease: The PREDIC-DIV Study
Brief Title: PREDICtors for Quality of Life After Sigmoidectomy for DIVerticular Disease
Acronym: PREDIC-DIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Städtisches Klinikum München GmbH (Other)
Responsible Party: Principal Investigator, Dr. Maximilian Sohn, Dr. med., Attending, Städtisches Klinikum München GmbH
Other Study IDs: PREDIC-DIV 1.0
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Diverticular Disease of Colon; Quality of Life
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The resected part of the bowel is histopathologically examinated and stored routinely for all patients (participants of the study as well as not participating patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify predictors for postoperative health related quality of life after elective sigmoidectomy for diverticular disease.

DETAILED DESCRIPTION:
According to current international guidelines, indications for surgical treatment of diverticular disease are inhomogeneous. To date, the measurement of pre- and postoperative quality of life (QoL) is underrepresented. To ensure an individually tailored therapeutical approach, and to avoid unnecessary surgery as well as the risk of a hazardous chronification of the disease, QoL importantly needs to be focused within the decisional process for the best treatment option. The aim of the PREDIC DIV-Study is, to identify predictors for a better postoperative quality of life in patients who undergo elective sigmoidectomy for diverticular disease. PREDIC DIV is a prospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* patients, scheduled for elective sigmoidectomy for diverticular disease (Indication: foregoing acute diverticulitis with pericolic or pelvic abscess >1cm, ongoing complaints after acute uncomplicated diverticulitis, recurrent uncomplicated disease (three or more diverticulitis episodes in combination with the patients wish for surgery), recurrent complicated disease (three or more diverticulitis episodes+complications: stenosis, fistula, chronic pain), urgent wish of patients for surgery after uncomplicated disease.
* Age >18 years
* ASA 1-3
* informed consent

Exclusion Criteria:

* Age <18 years
* ASA 4
* acute diverticulitis with free perforation
* acute or forgoing diverticular bleeding
* colorectal malignancies (current or foregoing)
* immunosuppression (corticoids > 20 mg prednisolon/d, status post transplant)
* advanced malignancy with systemic metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients > 18 years, matching to inclusion and exclusion criteria, who are scheduled for elective sigmoidectomy for diverticular disease
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative quality of life (QoL) after a follow up of six month: GI-Quality of Life Index | six month
  Quality of life will be assessed by use of the GI-Quality of Life Index

SECONDARY OUTCOMES:
Postoperative quality of life (QoL) after a follow up of six month: SF36 | six month
  Quality of life will be assessed by use of the SF36-questionnaire
Postoperative quality of life (QoL) after a follow up of six month: Visual analogue scale (VAS) | six month
  Quality of life will be assessed by use of a visual analogue scale (VAS). The scale ranges from 0 to 100 mm. 0 is the least desirable condition. 100 is the most desirable condition.
Quality of life after a follow up of 24 month: SF-36 | 24 month
  Quality of life will be assessed by use of SF36-questionnaire
Quality of life after a follow up of 24 month: GI-Quality of Life Index | 24 month
  Quality of life will be assessed by use GI-Quality of Life index-questionnaire
Quality of life after a follow up of 24 month: Visual analogue scale (VAS) | 24 month
  Quality of life will be assessed by use of a visual analogue scale (VAS). The scale ranges from 0 to 100 mm. 0 is the least desirable condition. 100 is the most desirable condition.
Peri- und postoperative morbidity | 30 days, 6 and 24 month
  Assessement by use of Clavien-Dindo-Classification
Mortality | 30 days, 6 and 24 month
  Mortality is defined as 30-days postoperative mortality and mortality in association to diverticulitis recurrency
Coexisting characteristics of irritable bowel syndrome (IBS) | 0, 6 and 24 month
  IBS-scoring will be performed pre- and postoperatively by use of ROME IV criteria
Subjective assessment of Diverticulitis severity | 0, 6 and 24 month
  Evaluation of the patients subjective estimate on disease severity by use of a visual analogue scale (VAS). The scale ranges from 0 to 100 mm. 0 is the least desirable condition (=most severe imaginable diverticulitis). 100 is the most desirable condition (=no diverticulitis).
Diverticulitis severity: Classification of Diverticular Disease | 1 day before surgery
  CT-scan based grading of diverticulitis in uncomplicated or complicated disease according to Classification of Diverticular Disease
Diverticulitis severity: Ambrossetti Classification | 1 day before surgery
  CT-scan based grading of diverticulitis in uncomplicated or complicated disease according to Ambrossetti Classification
Diverticulitis severity: Modified Hinchey Classification | 1 day before surgery
  CT-scan based grading of diverticulitis in uncomplicated or complicated disease according to Modified Hinchey Classification
Diverticulitis severity according to preoperative CT-scan | 1 day before surgery
  Evaluation for evidence of pericolic gas
Diverticulitis severity according to preoperative CT-scan | 1 day before surgery
  Evaluation for evidence of pericolic or pelvic abscess
Diverticulitis severity | 2 days after surgery
  histological grading of inflammation in the resected bowel (Grade 1-4)
Influence of guideline specific treatment on postoperative quality of life | 6 and 24 month
  Postoperative comparison of indication for surgery with given indications in relevant international Guidelines (German, US, Danish, GB, Italian, Dutch). Review of the association between a guideline-matching treatment and postoperative quality of life. Identification of the guideline, which potentially leads to the best achieved quality of life
Postoperative changes in fecal continence | 0, 6 and 24 month
  Pre- and postoperative results of Wexner-score
Postoperative changes in urinary continence | 0, 6 and 24 month
  Pre- and postoperative results of urinary distress inventory (UDI6)
Postoperative changes in male sexual function | 0, 6 and 24 month
  Assessment of male sexual function by use of International index of erectile function (IIEF)
Postoperative changes in female sexual function | 0, 6 and 24 month
  Assessment of female sexual function by use of Female Sexual Function Index (FSFI)
Preoperative fecal calprotectin | 1 day preoperative
  Measurement of fecal calprotectin preoperatively
Postoperative fecal calprotectin | 6 and 24 month
  Measurement of fecal calprotectin postoperatively
Morphological changes of the bowel wall | 1 day after surgery
  Analysis at the rectosigmoidal junction: overall thickness of the bowel wall
Morphological changes of the bowel wall: thickness of bowel wall | 1 day after surgery
  Analysis at the the rectosigmoidal junction: thickness of the muscular layer
Morphological changes of the bowel wall: Cells of Cajal | 1 day after surgery
  Analysis within the inflamed segment: amount of Cajal-cells in the bowel wall
Morphological changes of the bowel wall: Fibrosis | 1 day after surgery
  Analysis within the inflamed segment: Grade of fibrosis (1-4)
Cost analysis | baseline and 6 and 24 month
  Review of disease specific health cost by request at health insurance companies
Productivity analysis | baseline and 6 and 24 month
  Assessment of labour productivity by use of the Productivity Cost Questionnaire (iPCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Sohn, Dr. med., Study Director — Städtisches Klinikum München GmbH
Locations (1):
- Klinik für Allgemein- Viszeral-, Endokrine- und Minimalinvasive Chirurgie, Klinikum Bogenhausen, Städtisches Klinikum München GmbH, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Sohn M, Agha A, Iesalnieks I, Bremer S, Trum S, Di Cerbo F, Nerlich A, Lotz N, Klieser E, Hochrein A, Schredl P, Kalcheva D, Emmanuel K, Presl J. PREDICtors for health-related quality of life after elective sigmoidectomy for DIVerticular disease: the PREDIC-DIV study protocol of a prospective multicentric transnational observational study. BMJ Open. 2020 Mar 24;10(3):e034385. doi: 10.1136/bmjopen-2019-034385. PMID 32209628